CLINICAL TRIAL: NCT05733377
Title: Validation of a Non-invasive Image Technique for Studying Pregnant Women´s Lordosis. Relation Between Lordosis and Childbirth Outcome.
Brief Title: Non-invasive Imaging Technique for the Study of Lordosis in Pregnant Women and Its Relationship to Birth Outcome
Status: Recruiting | Type: Observational
Sponsor: University of Alcala (Other)
Collaborators: Hospital Universitario de Fuenlabrada (Other)
Responsible Party: Principal Investigator, Susana Nunez Nagy, Professor, PhD, University of Alcala
Other Study IDs: Pregnant women´s lordosis
Record Dates: First submitted 2023-01-30; First posted 2023-02-17 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Pregnancy Outcome; Biomechanics; Back Disorder; Diagnostic Imaging; Biomedical Technology

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pregnant: Pregnant >36 weeks gestation, 20 to 40 years old, without significant lumbar pathology, or intense labor pain, or percentile p>97 or <p3, or with a result of delivery-cesarean section due to risk of loss of fetal well-being
  Interventions: Diagnostic Test: Arrow Test; Diagnostic Test: Angle measurement by imaging device

INTERVENTIONS:
Diagnostic Test: Arrow Test — It consists of taking the widest measurement between the rope of a plumb bob on her upper and lower back.
Diagnostic Test: Angle measurement by imaging device — First, three anatomical landmarks are located, and a sticker is placed on each of them: the 12th thoracic vertebra at its intersection with the midline descending from the axilla, the greater trochanter, and the anterior superior iliac spine. After this, the woman will be asked to stand in a normal position facing forward with her hands crossed over her shoulders, and a picture will be taken and pixelated with anything that could identify her. The angle formed by the three stickers will be measured with this image and the software.

SUMMARY:
The study consists of collecting measurement data of the rachis in pregnant women and the subsequent outcome of her delivery.

This will make it possible to validate a non-invasive imaging technique through software that can be used to study this anatomical curve proposing a new measurement method for the angle of lordosis.

Finally, with the research data, the investigators will try to find a correlation between these variables (angle of lordosis and delivery outcome.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women between 20 and 40 years old with a low-risk pregnancy

Exclusion Criteria:

* Pregnant women under 20 years and over 40 years of age or with a significant lumbar pathology or with a very high-risk pregnancy or with IMC >35

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Pregnant women are being monitored by the Fuenlabrada Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 122 (Estimated)
Dates: Start 2022-07-15 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Lordosis angle using an app | 2025
  Differentiation between lordosis, hyperlordosis and lumbar rectification

SECONDARY OUTCOMES:
Lordosis angle by means of arrow test | 2025
  Differentiation between lordosis, hyperlordosis and lumbar rectification.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alcalá, Alcalá de Henares, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No